CLINICAL TRIAL: NCT00438581
Title: Phase II Non-Randomized Study Combining Yttrium 90 Ibritumomab Tiuxetan (Zevalin) With High-Dose Chemotherapy Prior to Autologous Stem Cell Transplantation in Patients With Relapsed, Refractory, or Transformed Non-Hodgkin's Lymphoma
Brief Title: Study Combining Zevalin With High-Dose Chemotherapy Prior to Autologous StemCell Transplant in Patients With Relapsed, Refractory, or Transformed Non-Hodgkin's Lymphoma
Acronym: Zevalin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMA-05-017-ZEV
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Zevalin; Autologous one Marrow Transplant; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan

INTERVENTIONS:
Drug: Yttrium 90 Ibritumomab Tiuxetan ( Zevalin )

SUMMARY:
This aim of this study to evaluate the safety and efficacy of combining a single course of Yttrium 90 Ibritumomab Tiuxetan, a radiolabeled monoclonal antibody ( Zevalin ), with high-dose BEAM chemotherapy and autologous peripheral stem cell transplantation in patients with relapsed, refractory, or transformed Non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Relapse rates after chemotherapy for relapsed, refractory or transformed Non-Hodgkin's lymphoma (NHL)remain very high. NHL is a radiosensitive tumor. We hypothesize that targeted radioimmunotherapy combined with high-dose chemotherapy may increase response and survival rates in a safe and reliable manner.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 to <=70 years
2. Relapsed or refractory Stage III or IV, grade 1,2, or 3 Follicular Lymphoma or transformed follicular lymphoma, mantle cell lymphoma, marginal zone lymphoma, Waldenstrom's macroglobulinemia, or diffuse large B-Cell lymphoma as defined by the WHO and:

   * Expressing the CD 20 antigen
   * ECOG performance 0-2
   * Written informed consent
3. Prior collection of at least 2.5x10^6 CD34-positive peripheral blood stem cells/kg.

Exclusion Criteria:

1. Abnormal renal function (Creatinine >2.5x upper limit of normal (ULN)
2. Abnormal hepatic function (Bilirubin >2xULN, ALT/AST >3x ULN)
3. Cardiac ejection fraction <40%
4. Severe defects in pulmonary function tests (DLCO<70% predicted, FEV1, FVC<60% predicted) or receiving continuous oxygen
5. A history of human anti-mouse antibodies (HAMA) or known type 1 hypersensitivity or anaphylactic proteins to any component of the Zevalin therapy.
6. Female patients who are pregnant or breast feeding, and adults of reproductive potential who are not employing an effective method of birth control during study treatment
7. Prior radiotherapy to >25% of the bone marrow or >20 Gy to critical organ (lung, liver, kidney, spinal cord).
8. CNS lymphoma
9. Ongoing infection
10. Prior treatment with radioimmunotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-03

PRIMARY OUTCOMES:
Overall response rate

SECONDARY OUTCOMES:
Survival Data, adverse events, molecular response

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Galal, MD, Principal Investigator — McGill University Health Center, Royal Victoria Hospital
Locations (1):
- McGill University Health Center, Royal Victoria Hospital, Montreal, Quebec, Canada